CLINICAL TRIAL: NCT03056924
Title: Immunogenicity of Influenza, Pneumococcal and Hepatitis B Vaccines in Inflammatory Bowel Disease Patients Treated With Vedolizumab
Brief Title: Immunogenicity of Influenza, Pneumococcal and Hepatitis B Vaccines in IBD Patients Treated With Vedolizumab
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-35669
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine; Influenza Vaccines; Afluria; Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Vedolizumab monotherapy: IBD patients on vedolizumab monotherapy, all patients will be treated with the standard vedolizumab dosing regimen of 300 mg infusions at 8 week intervals and receive Pneumococcal Pneumonia vaccine and/or Influenza vaccine and/or Hepatitis B vaccine.
  Interventions: Biological: Pneumococcal Pneumonia vaccine; Biological: Influenza vaccine; Biological: Hepatitis B vaccine
- vedolizumab + immunomodulator: IBD patients receiving combination treatment with vedolizumab and concomitant immunomodulator therapy (methotrexate, azathioprine, or 6-mercaptopurine), will be treated with the standard vedolizumab dosing regimen of 300 mg infusions at 8 week intervals and/or receive Pneumococcal Pneumonia vaccine and/or Influenza vaccine and/or Hepatitis B vaccine.
  Interventions: Biological: Pneumococcal Pneumonia vaccine; Biological: Influenza vaccine; Biological: Hepatitis B vaccine
- biologic + immunomodulator: IBD patients on other biologic therapy (infliximab, adalimumab, certolizumab, golimumab, ustekinumab) with concomitant immunomodulator therapy (methotrexate, azathioprine, or 6-mercaptopurine) and receivePneumococcal Pneumonia vaccine and/or Influenza vaccine and/or Hepatitis B vaccine.
  Interventions: Biological: Pneumococcal Pneumonia vaccine; Biological: Influenza vaccine; Biological: Hepatitis B vaccine
- non-immunosuppressive therapy: IBD patients not taking any immunosuppressive therapy (these patients may be taking oral or topical 5-aminosalicylates) and recive Pneumococcal Pneumonia vaccine and/or Influenza vaccine and/or Hepatitis B vaccine.
  Interventions: Biological: Pneumococcal Pneumonia vaccine; Biological: Influenza vaccine; Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Pneumococcal Pneumonia vaccine — Vaccination for pneumococcal pneumonia will be carried out with either the PSV-23 (Pneumovax, Merck, Whitehouse Station, NJ) or the PCV-13 (Prevnar 13, Pfizer, Philadelphia, PA). Either vaccine is administered in a single dose of 0.5 mL intramuscularly.
  Other Names: PSV-23 (Pneumovax, Merck, Whitehouse Station, NJ); PCV-13 (Prevnar 13, Pfizer, Philadelphia, PA).
Biological: Influenza vaccine — Influenza vaccination will be carried out with the 2017-2018 trivalent component vaccine (Afluria, Seqirus USA Inc., King of Prussia, PA) or for patients over 65 years of age (Fluzone, Sanofi Pasteur, Swiftwater, PA). Both of these vaccines are administered in a single dose of 0.5 mL intramuscularly.
  Other Names: Afluria; Fluzone
Biological: Hepatitis B vaccine — Hepatitis B vaccination with be carried out with a single antigen, recombinant hepatitis B vaccine (Energix B, GlaxoSmithKline, Research Triangle Park, NC). This vaccine is administered in a three dose series with 1.0 mL given intramuscularly at 0, 1, and 6 months. For patients receiving a booster, a single intramuscular dose of 1.0 mL will be given.
  Other Names: Energix B

SUMMARY:
Patients with Crohn's disease (CD) and ulcerative colitis (UC) are often treated with medications that suppress the immune system. These patients are therefore at increased risk for developing infections, such as influenza, pneumonia, and hepatitis B, which may be prevented by vaccination. While awareness is increasing among gastroenterologists of the importance of vaccinations in the IBD patient, there continues to be some question of the effectiveness of vaccination in immunosuppressed patients. It has been previously shown that patients on immunosuppressive therapy with certain biologic medications (the TNF-blockers: infliximab and adalimumab) had an impaired immune response to vaccination as compared to healthy controls, as the mechanism of immunosuppression for these agents is systemic. Vedolizumab, a biologic medication for CD and UC approved in May 2014, targets the α4β7 integrin, a key component of gut immunity, and as such it has been hypothesized that with this agent effects are gut specific. There is limited data that suggests that in healthy patients given vedolizumab do not have an altered response to parentally administered vaccines, however there are no studies in the CD and UC population describing this. Additionally, IBD patients treated with vedolizumab are frequently also on concomitant therapy with an immunomodulator (6-mercaptopurine, azathioprine, or methotrexate), and these patients ability to mount an immune response has not been demonstrated.

DETAILED DESCRIPTION:
The purpose of this study is to determine immune response rates to (a) influenza, (b) pneumococcal, and (c) hepatitis B vaccines in IBD patients receiving vedolizumab therapy compared to patients on other therapies for IBD.

Four study groups will be established -- 1. Group A - IBD patients on vedolizumab monotherapy. 2. Group B - IBD patients receiving combination treatment with vedolizumab and concomitant immunomodulator therapt (methotrexate, azathioprine, or 6-mercaptopurine). 3. Group C - IBD patients on other biologic therapy (infliximab, adalimumab, certolizumab, golimumab, and ustekinumab). 4. Group D - IBD patients not taking any immunosuppressive therapy. Patients in all groups should have been on stable treatment for IBD for at least three months.

For each of the four vaccines included in this study (influenza, PCV-13, PSV-23, hepatitis B), a total of 220 samples will be collected. Given that more than one of these vaccines may be clinically indicated for an individual patient, a single patient may receive more than one vaccine, and therefore can be included in the immune response analysis for each vaccine they receive.

Once the subject has signed consent and enrolled in the study, the following procedures will take place:

Baseline/enrollment visit: The subject will have a comprehensive medical history and physical exam performed at their baseline clinic visit. During this visit they will also fill out the 10 question IBD quality of life questionnaire, a baseline serum sample will be obtained, and then receive the vaccine(s) indicated based on their vaccination history. These vaccines include, for pneumococcal pneumonia - PSV-23 and PCV-13 (both given as a single dose of 0.5 mL intramuscularly in the deltoid region of the upper arm), for influenza - Afluria or Fluzone for patients over 65 year of ago (both given as a single dose of 0.5 mL intramuscularly in the deltoid region of the upper arm), and for hepatitis B - Energix (administered in a three dose series with 1.0 mL given at 0, 1, and 6 months, or for patients receiving a booster a single intramuscular dose of 1.0 mL will be given). Subjects will be instructed to call the study team for any concerns or any development of fever, chills, rash or other concerning symptom.

Follow up phone call: Subjects will receive a follow-up phone call 2 weeks after vaccination to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physicians.

Follow up visit: At 3-4 weeks after vaccination, patients will have a visit where serum will again be obtained. Patients will also be asked about any adverse events such as fevers or vaccine reactions, as well as complete the 10 question IBD quality of life questionnaire (IBDQ).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-75 with IBD (diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria) receiving care at Boston Medical Center, Center for Digestive Disorders.
2. Patients receiving one of the following treatments for their IBD - vedolizumab monotherapy, combination treatment with vedolizumab and concomitant immunomodulator therapy (methotrexate, azathioprine, or 6-mercaptopurine), combination treatment with a TNF inhibitor and concomitant immunomodulator therapy (methotrexate, azathioprine, or 6-mercaptopurine), or no immunosuppressive therapy (these patients may be taking oral or topical 5-aminosalicylates). Patients in all groups should have been on stable treatment for IBD for at least three months.

Exclusion Criteria:

1. Any patients with prior vaccination with the intended vaccine, with the exception of those receiving a hepatitis B booster.
2. Any patient with an allergy to the vaccine components.
3. Patients who cannot provide informed consent.
4. Patients who are being administered any non-licensed or experimental immunomodulators
5. Patients taking steroids orally or intravenously (more than 20mg prednisone or equivalent dose of other corticosteroids) for at least 10 days, within the 30 days prior to vaccination.
6. Patients who have received immunoglobulin therapy or blood products within the past one month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-75 with IBD (diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria) receiving care at Boston Medical Center, Center for Digestive Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of immune seroconversion after influenza, pneumococcal, or hepatitis B vaccine among the four groups of patients | baseline and 3 - 4 weeks
  The primary outcome is percent change in IgG titer from baseline to 3 weeks post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmeel K Wasan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided